CLINICAL TRIAL: NCT04499716
Title: Quadriblock Versus "IPACK + Femoral Triangle Block + Obturator Nerve Block" in Total Knee Arthroplasty: a Randomized Controlled Clinical Trial
Brief Title: Quadriblock Versus "IPACK + Femoral Triangle Block + Obturator Nerve Block" in Total Knee Arthroplasty
Acronym: QuITO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Medipole Garonne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020/04
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2020-07

CONDITIONS: Primary Total Knee Arthroplasty
Keywords: Knee arthroplasty, Regional anesthesia, Ropivacaine, Postoperative analgesia, Pain management, Opioids
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: ITO group (Active Comparator): Arm 1: IPACK combined with femoral triangle and obturator nerve blocks
  Interventions: Procedure: IPACK; Procedure: Femoral triangle block; Procedure: Obturator nerve block
- Arm 2 : Quadri-block group (Experimental): Arm 2 : Femoral, sciatic, obturator and lateral femoral cutaneous nerve blocks
  Interventions: Procedure: Obturator nerve block; Procedure: Femoral nerve block; Procedure: Sciatic nerve block; Procedure: Lateral femoral cutaneous nerve block

INTERVENTIONS:
Procedure: IPACK — 25 milliliters of ropivacaine 0.3% will be injected between popliteal artery and femur.
  Arms: Arm 1: ITO group
Procedure: Femoral triangle block — 25 milliliters of ropivacaine 0.3% will be injected on the lateral side of the femoral artery at the distal part of the femoral triangle.
  Arms: Arm 1: ITO group
Procedure: Obturator nerve block — 20 milliliters of ropivacaine 0.3% will be injected between the adductor magnus and adductor brevis muscles and between the adductor brevis muscle the pectineus.
Procedure: Femoral nerve block — 20 milliliters of ropivacaine 0.3% will be injected in supine position under the fascia iliaca lateral to the femoral artery.
  Arms: Arm 2 : Quadri-block group
Procedure: Sciatic nerve block — 25 milliliters of ropivacaine 0.3% will be injected in prone position in the subgluteal space by lateral approach.
  Arms: Arm 2 : Quadri-block group
Procedure: Lateral femoral cutaneous nerve block — 5 milliliters of ropivacaine 0.3% will be injected laterally to the sartorius muscle.
  Arms: Arm 2 : Quadri-block group

SUMMARY:
Total knee arthroplasty (TKA) is one of the most common orthopedic surgical procedure and is associated with severe pain in the immediate postoperative period, thus limiting early recovery.

Postoperative pain management requires multimodal analgesia, combining drugs and injection of a local anesthetic (LA). For optimal pain management, several peripheral nerve blocks should be associated. Thus, a recent study shows that the combination of IPACK, femoral triangle and obturator nerve blocks (ITO blocks) provides an effective pain control after TKA.

The hypothesis of this study is that a quadruple nerve block combining femoral, sciatic, obturator and lateral femoral cutaneous nerve blocks (quadri-block) could improve analgesia after TKA.

The main objective of this monocenter, prospective, randomized, open-label, controlled trial is to assess the effect of quadri-block on morphine consumption after TKA compared to ITO blocks.

DETAILED DESCRIPTION:
In the pre-anaesthesia room, after the implementation of classical monitoring with an oxygen mask and a peripheral venous catheter, all patients will receive an antibioprophylaxis according to SFAR (French Society of Anesthesia & Intensive Care Medecine) recommendations and injection of 10 mg of IV dexamethasone.

The patients will be then randomized in 2 groups:

* ITO group (usual technique): IPACK combined to femoral triangle and obturator nerve blocks
* Quadriblock group (experimental technique): femoral, sciatic, obturator and lateral femoral cutaneous nerve blocks.

An experienced anesthetist will perform ultrasound-guided blocks 30 minutes before surgery with ropivacaine 0.3%, total volume of 70 ml.

In the operating room, general anesthesia will be induced by intravenous ketamine (0.4 mg/kg) and propofol (3 mg/kg). Anesthesia will be maintained with propofol.

Postoperative analgesia protocol :

* Multimodal analgesia will be instituted from the end of the surgery by the administration of paracetamol (1 g) and ketoprofen (100 mg).
* In post-anesthesia care unit (PACU): oxynorm titration if VRS (pain score) >3 according to the centre's usual care.
* In ward: systematic per os analgesia with paracetamol (1 g, 4 times a day) and ibuprofen (400 mg, 3 times a day); oxynorm (10 mg, lockout interval: 4 h) if VRS (pain score) >3.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* Primary total knee arthroplasty
* Consent for participation,
* Affiliation to a social security system

Exclusion Criteria:

* Preoperative morphine use
* Chronic pain syndrome
* Contraindication to any drugs used in the protocol (paracetamol, ketoprofen, oxynorm, propofol, ketamine, ropivacaine)
* Valgus > 9°
* Pregnant or breastfeeding women
* Patients under protection of the adults (guardianship, curators or safeguard of justice)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia, defined by the morphine consumption in the first 48 hours post-surgery. | 48 hours
  Total amount of oxynorm (mg) administered during the first 48 hours post-surgery.

SECONDARY OUTCOMES:
Postoperative pain: Verbal Rating Scale (VRS) | 48 hours
  Pain will be assessed every 6 hours using a Verbal Rating Scale (VRS) ranging from 0 to 10 (0=no pain, 10=worst possible pain).
Oxynorm consumption in the first 24 hours post-surgery | 24 hours
  Total amount of oxynorm (mg) administered during the first 24 hours post-surgery.
Ability to walk | 48 hours
  0: unable to get up; 1: able to get up but not to walk; 2: walk <50 m; 3: walk > 50 m
Quadricep mobilization | 48 hours
  0: paralysis; 1: paresis, 2: normal contraction
Foot elevator muscle mobilization | 48 hours
  0: paralysis; 1: paresis; 2: normal contraction
Side effects of opioids | 48 hours
  Collect side effects associated with oxynorm : nausea or vomiting, drowsiness, constipation, urinary retention, itching, disorientation.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Médipôle Garonne, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marty P, Chassery C, Rontes O, Vuillaume C, Basset B, Merouani M, Marquis C, De Lussy A, Ferre F, Naudin C, Joshi GP, Delbos A. Combined proximal or distal nerve blocks for postoperative analgesia after total knee arthroplasty: a randomised controlled trial. Br J Anaesth. 2022 Sep;129(3):427-434. doi: 10.1016/j.bja.2022.05.024. Epub 2022 Jun 28. PMID 35773028